CLINICAL TRIAL: NCT06532526
Title: Assessment of the Effects of Bio-active Desensitizing Materials on the Bleaching Efficacy and Reduction of Tooth Sensitivity Caused by Vital In-office Bleaching: A Randomized Controlled Clinical Trial
Brief Title: Effects of Bio-active Desensitizer on Reduction of Tooth Sensitivity Caused by In-office Bleaching.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Principal Investigator, Ghada Maghaireh, Dr., King Abdullah University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 886-2023
Record Dates: First submitted 2024-07-25; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Tooth Discoloration
Keywords: Sensitivity; Bio-active desensitizer; in-office bleaching
MeSH Terms: conditions — Tooth Discoloration; Hypersensitivity | interventions — Gels; Sodium Fluoride

STUDY DESIGN:
Intervention Model Description: The study will be a double blinded (Patient and evaluator) randomized clinical trial with a sample size of 51, 17 participants for each group (n=17).
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants as well as the evaluators will be informed about the nature and objectives of the study; however, they will not be informed what desensitizing material they would receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First group (Active Comparator): Predicat Bioactive desensitizer
  Interventions: Other: Predicta® Bioactive Desensitizer (PBD, PARKELL, EDGEWOOD, NY, USA)
- Second group (Active Comparator): Gel with 1.23% sodium fluoride
  Interventions: Other: Gel with 1.23% sodium fluoride (EAZIGEL, VERICOM CO., LTD. SOUTH KOREA)
- Third group (Placebo Comparator): Placebo gel
  Interventions: Other: Placebo gel without any active ingredients.

INTERVENTIONS:
Other: Predicta® Bioactive Desensitizer (PBD, PARKELL, EDGEWOOD, NY, USA) — A bioactive desensitizer gel that applied on teeth to reduce tooth sensitivity associated with dental bleaching.
  Arms: First group
Other: Gel with 1.23% sodium fluoride (EAZIGEL, VERICOM CO., LTD. SOUTH KOREA) — Fluoride gel that applied on the teeth to reduce tooth sensitivity
  Arms: Second group
Other: Placebo gel without any active ingredients. — Water-based glycerin gel is used as the Placebo gel without active ingredients
  Arms: Third group

SUMMARY:
The main aim of this randomized controlled clinical trial is to evaluate the efficacy of a bioactive glass desensitizer in reducing tooth sensitivity associated with in-office vital tooth bleaching. In addition, this study aims to compare the effectiveness of the bioactive glass desensitizer with that of a fluoride gel and a gel without desensitizing agent with regard to incidence, intensity, and duration of tooth sensitivity and, finally, to investigate how these agents affect tooth-shade following in-office bleaching. The hypothesis of the study is: There will be no difference in the effect of a bio-active glass desensitizer on tooth sensitivity associated with vital in-office tooth bleaching compared to a fluoride gel and the bio-active glass desensitizer has no effect on the bleaching efficacy.

DETAILED DESCRIPTION:
The participants will be informed about the nature and objectives of the study; however, they will not be informed what desensitizing material they would receive. The study will be a double blinded (Patient and evaluator) randomized clinical trial with a sample size of 51, 17 participants for each group (n=17). Bleaching process: A lip and cheek retractor will be placed. The gingival tissues from the right first molar to the left first molar will be isolated using a light-cured resin dam to prevent the whitening gel from coming into contact with the gingival tissue. Participants' lips will be painted with Vaseline, and protective eyewear will be used. To aid in the isolation process, a plastic suction tip with high suction power will be used. Opalescence Boost in Office Whitening Gel, 40% Hydrogen Peroxide bleaching material (Ultradent Products, South Jordan, UT, USA) will be applied directly on the labial tooth surface from the right first premolar to the left first premolar. A total of three (20-minute) applications will be completed in each bleaching session. Participants will undergo 2 bleaching sessions with one-week interval. Participants will be scheduled for lower arch whitening after 14 days.

Application of the desensitizer: The participants will be assigned randomly to three study groups. The first group will receive a bio active desensitizer, the second group will receive a fluoride gel and the third group will receive a placebo gel without a desensitizer (Table 2). A small amount of the gel assigned for each participant will be applied directly on the labial surface of each tooth and left undisturbed for three minutes; care will be taken to cover the entire labial surface, and the gel will be carried interproximally as much as possible.

Shade evaluation: Teeth shade will be evaluated subjectively and objectively. Subjectively it will be evaluated using VITA classical shade guide which has 16 tabs ranging from B1 (lightest value) to C4 (darkest value) by matching the color with the middle third of the maxillary anterior teeth. One evaluator will record the shade of the participants' teeth at baseline (before whitening), directly after bleaching, and at days 3, 7, and 14 days follow up periods. Photographs will be taken using a digital camera immediately after the whitening and at each shade evaluation to document results. Also teeth shade will be evaluated objectively using VITA easy shade spectrophotometer (VITA Easyshade V; VITA Zahnfabrik, Bad Säckingen, Germany). The tooth must be well hydrated before analyzing the tooth color. The shade of the teeth in VITA classical A1-D4 and VITA 3D-MASTER shades will be instantly measured and displayed on the screen. One evaluator will record the shade of the teeth and the shade will be recorded at baseline, immediately after bleaching and at 3, 7 and 14 days follow up periods. Sensitivity Evaluation: Post-bleaching sensitivity will be evaluated by relying on patient's feeling of pain.

Sensitivity evaluation: All participants will be given a sensitivity sheet to record the post-whitening sensitivity of the whitened teeth on daily basis up to 14 days according to the visual analog scale of pain (VAS). The participants will be asked to record the stimulus that caused sensitivity, including hot, cold, or other. The duration of pain, whether seconds, minutes, or hours, will be recorded for the 14-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* At least eight maxillary anterior teeth present.
* Age between 18 and 30 years Smokers
* The selected teeth has a mean shade of C2 or darker (Vitapan Classical, Vita-Zahnfabrik, Sa¨ckingen, Germany)
* Good general and oral health (no visible plaque or gingivitis)
* No restorations or carious lesions on the buccal surfaces of the anterior teeth to be whitened
* No history of tooth sensitivity
* No use of a desensitizing agent or desensitizing toothpaste in the past six months

Exclusion Criteria:

* Active caries and/or periodontal diseases (gingivitis and recession) or wasting diseases
* Smokers
* Pregnant/lactating women
* Patients who have bleached their teeth previously
* No schedule availability

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Tooth sensitivity associated with vital in-office tooth bleaching | Assess sensitivity during the bleaching, 1 hour after bleaching, 1 day, 2 days, 7 days and 14 days after bleaching.
  Tooth sensitivity associated with vital in-office tooth bleaching using the the five-point Numeric Rating Scale (NRS):
  0: No sensitivity
  1. Mild sensitivity,
  2. Moderate sensitivity
  3. Considerable sensitivity
  4. Severe sensitivity Also, sensitivity will be evaluated using the visual analog scale of pain (VAS). The VAS is a horizontal line containing 10 numbers from 0 to 10; zero indicates no pain and 10 indicates the worst pain. Participants will be asked to mark the number that indicated their level of pain. The participants will be asked to record the stimulus that caused sensitivity, including hot, cold, or other. The duration of pain, whether seconds, minutes, or hours, will be recorded for the 14-day follow-up period. For descriptive analysis purposes, the intensity results will be categorized according to the following scale: 0 = none, 1-3 = mild, 4-6 = moderate, and 7-10 = severe.

SECONDARY OUTCOMES:
Efficacy of bleaching | Evaluate teeth shade subjectively and objectively after the removal of isolation and after 14 days of bleaching.
  Lightening of the teeth shade with in-office tooth bleaching. Subjectively it will be evaluated using VITA classical shade guide which has 16 tabs ranging from B1 (lightest value) to C4 (darkest value) by matching the color with the middle third of the maxillary anterior teeth. One evaluator will record the shade of the participants' teeth at baseline (before whitening), directly after bleaching, and at days 3, 7, and 14 days follow up periods. Photographs will be taken using a digital camera immediately after the whitening and at each shade evaluation to document results. Also, teeth shade will be evaluated objectively using VITA easy shade spectrophotometer (VITA Easyshade V; VITA Zahnfabrik, Bad Säckingen, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A Maghaireh, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maghaireh GA, Alzraikat H, Altarazi MY. Effects of a bioactive desensitizing material on in-office bleaching-induced tooth sensitivity: A randomized double-blind controlled trial. J Dent. 2026 Jan 1;166:106326. doi: 10.1016/j.jdent.2025.106326. Online ahead of print. PMID 41483835